CLINICAL TRIAL: NCT06591546
Title: Telescoping Nail Osteosynthesis in Management of Osteogenesis Imperfecta in Growing Child
Brief Title: Telescoping Nail in Osteogenesis Imperfecta
Acronym: Telescoping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Tarek Ismail Alkady Mohammed, Assistant lecturer at Al-Azhar university Assuit, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNOMOIGC
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteogenesis
Keywords: Osteogenesis imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Intervention Model Description: Growing child (3-12 ys) Bony deformities with other symptoms and signs of OI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telescoping nail (Experimental): The implant used in this study is Fassier Duval type of telescoping nail.
  The Fassier-Duval rod has certain advantages:
  the design is dedicated to minimally invasive, ideally percutaneous, approaches sparing joint cartilage at implant positioning and removal. This reduces the risk of delayed growth and infection, with lower scar impact; instrumentation is much better than the very basic Dubow-Bailey instrumentation; maximum diameter is greater: 6.4 mm, compared to 5 mm for Bailey-Dubow; The length of the female part can be adapted, including intraoperatively. Precutting according to the surgeon's measurement can be adjusted intraoperatively with a dedicated circular saw with a diamond disc.
  Interventions: Device: Telescoping nail

INTERVENTIONS:
Device: Telescoping nail — The implant used in this study is Fassier Duval type of telescoping nail.
  The Fassier-Duval rod has certain advantages:
  the design is dedicated to minimally invasive, ideally percutaneous, approaches sparing joint cartilage at implant positioning and removal. This reduces the risk of delayed growth and infection, with lower scar impact; instrumentation is much better than the very basic Dubow-Bailey instrumentation; maximum diameter is greater: 6.4 mm, compared to 5 mm for Bailey-Dubow; The length of the female part can be adapted, including intraoperatively. Precutting according to the surgeon's measurement can be adjusted intraoperatively with a dedicated circular saw with a diamond disc.

SUMMARY:
Osteogenesis Imperfecta (OI) is an autosomal dominant disorder that mainly affects the bones. Bones break easily. The severity may be mild to severe.

OI includes a blue tinge to the sclera of the eye, short height, loose joints, hearing loss, breathing problems and problems with the teeth. Complications may include cervical and aortic artery dissection.

Telescoping Nail Osteosynthesis:

The necessity for such treatment is given by the rapidly evolving anterior bowing (sometimes associated with rotation) and the increasing incidence of bone fracturing after cast removal. The decision to choose Sheffield-Millard osteotomies is based on the more than 20° angulation and the narrow medullar channel that makes reaming the only solution for passing the rod. Sometimes, in very severe cases, when the distance between the epiphysis gets smaller as the bone gets more and more bowed, it is imperative to do a shorting of the segment so that the soft tissues are not put in excessive tension after alignment.

Until the development of this technique, doctors used Kirschnerwire ,Kuntscher nails , Rush nails , Ender nails and most recently, elastic nailing . All the techniques had good short-term results, with good bone alignment and prevention of the refracturing of the bone. However, the biggest problem with these materials was that the patients outgrew them very fast, and problems like secondary bowing and refracturing appeared.

The aim of this study is the evaluation of the management of skeletal deformities in growing children with OI with telescoping nails.

This cross-sectional study was conducted. Twenty patients were included in this study operated at Alazhar University Hospital Assuit. The duration of the study ranged from 24-36 months.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is an autosomal dominant or recessive connective tissue disorder caused by the deficiency of Type I collagen production associated with the deficiency of collagen Type I alpha 1 chain and collagen Type I alpha 2 chain. This disease causes problems in all tissues that contain Type 1 collagen. In addition to many systemic problems such as blue sclera, otosclerosis, cardiac diseases, elasticity in the joint and thinning of the fascia, it also causes the loss of the normal ossification of the endochondral bone. This results in easily fragile bones. Although recurrent fractures show spontaneous healing traits, they lead to increased deformities developing with age . (24).

Osteogenesis Imperfecta (OI) is a hereditary condition affecting approximately 1 in 20,000 births with eleven recognized types of illness each one with its characteristics. Children with OI have low bone mass together with poor structural value, so, these two problems lead to recurrent fractures, varying degrees of short stature and progressive deformities of the limb and of the whole body in general. Severity ranges from those mildly affected individuals (Type 1) who have minimal bone deformity, near normal stature, blue sclerae and variable hearing loss, to those who are lethally affected with multiple fractures both in utero and in the first month of life that lead to respiratory failure and death . (25).

On top of all these problems, the most important and dramatic one regards the bone system, and, the way it manifests itself is by brittleness of the bones that leads to more and more fractures as the child grows, the peak being in the first years after the walking age, that is about one year and 2 months to 1 year and 6 months. In all the cases this is the point when something must be done immediately because the prognosis goes from worse to worse as time goes by when the child grows and begins to walk, thus limiting the childs capacity for a normal life. The main drawback of not doing something to stabilize the bones and reinforce them is the development of progressive deformities of the bone that add up more stress on the child, parents and eventually on the medical staff because surgery gets riskier and more complex . (35).

In OI cases, osteosynthesis performed with intramedullary nailing is the gold standard for surgical treatment to be administered following fracture and deformity. Intramedullary nailing, together with its corrective effect on deformity, is also effective in preventing recurrent fractures. Intramedullary nailing should be performed in a way that does not hinder the growth of children and should minimize the need for repetitive surgery as the child grows . (36).

There are a limited number of intramedullary nail types designed for this purpose and research is underway for the ideal nail. Today, telescopic nails with elastic or extendable features are frequently resorted. With elastic nails, there was a problem of migration (retraction) over time, while the problem encountered in telescopic nails was the need to open the joint (arthrotomy) during fixation to prevent migration, which posed another challenge . (85).

The main aim of this study was to evaluate the management of skeletal deformities in growing children with OI with telescoping nail.

This case series study was conducted. Twenty patients were included in this study operated at Alazhar University Hospital Assuit. The duration of the study ranged from 24-36 months.

The main results of this study were as following:

As regards the demographic data of the studied group. Age was ranged between 3 - 13 years with a mean value of 7.65±2.907 years. More than half were female (56.0%).

Our results were in agreement with study of Sterian et al.,(87) as they reported that the study group consisted of 12 patients both males and females, with ages ranging from 2 years and 3 months to 12 years, with the male: female ratio of 1:2.

However, in the study of Persiani et al.,(101) they selected 36 patients with OI type 3 (15 females and 21 males), aged between 2 and 10 years old to conduct their study.

The present study showed that as regards the operated bone of the studied group. The majority had the femur as an operated bone and the half of patients had the operated bone on the right side.

Our results were supported by study of Günay et al. (103) as they reported that six of the nails were applied to the tibia, and 14 to the femur.

Osteogenesis imperfecta (OI) is a genetic disorder of connective tissue that, in 70% of individuals, is caused by mutations of one of two genes (COL1A1 and COL1A2) that encode for the type I collagen chains. The major clinical features of OI are bone fragility, osteopenia, varying degrees of short stature, and progressive skeletal deformity. Other clinical features include joint hypermobility, hypotonia, and delayed or arrested developmental milestones in the more severely affected children. Its reported incidence ranges from approximately 1 in 10,000 to 1 in 20,000 births . (25).

The current study showed that as regard the family history of consanguinity of the studied sample show that 14(70%) had a family history of consanguinity.

In the study in our hands, as regards the past history of operations of the studied sample show that 10(50%) had Past history of operations and more than half of them with IM flexible nail (60%).

In a case reported held by Sterian et al.(87), they dealt with the case of a patient diagnosed with Osteogenesis Imperfecta at the age of 3 months. By that time, he already suffered 3 left femur fractures, one of which was at the age of 7 months, in utero, being accidentally diagnosed during a checkup the mother had at that time. Until the age of 4 years, the patient suffered 8 fractures of the lower limbs, all of them located at the level of the femurs, evenly distributed amongst right and left. Until that age, the treatment was done solely orthopedically. No cast immobilization and surgery were undergone to correct the bone deformity that developed or any kind of osteosynthesis.

Also, Popkov, (104)revealed that the past medical history was significant for multiple fractures managed conservatively. The diagnosis of OI type VIII had been established using a targeted next-generation sequencing approach.

Furthermore, Sterian et al.,(87) demonstrated that all of their studied cases came to the hospital late, after walking, after several fractures occurred and the only treatment, they underwent was prolonged cast immobilization that caused rapid bone demineralization, axial deformations of the affected bones, increased number of fractures and eventually loss of ambulation. The only treatment for these cases was surgery and the method proposed was Sofield-Miller corrective osteotomies and Fassier-Duval telescopic nail osteosynthesis. Prior to the surgical intervention, patients had a bisphosphonate treatment for 7 days.

Bisphosphonates (BP) is an analog of pyrophosphate, which slows down bone resorption and inhibits the function of osteoclasts. Numerous studies have shown that BPs increase BMD, improve bone architecture, prevent the progression of long bone deformities, restore the size and shape of vertebrae after compression fractures, foster growth, and increase mobility in children with OI. In several works, BP has been shown to reduce the frequency of long bone fractures. BP has been proven to be more effective in children than in adults. BPs do not affect the course of scoliosis because they do not reduce joint hyper-elasticity, which is the main cause of scoliosis. (62).

OI patients are administered with BP both intravenously and orally. The advantages of intravenous administration are the possibility of dose titration, better bioavailability, and the absence of side effects in the gastrointestinal tract. However, comparative studies did not show a significant difference in the effectiveness of intravenous and oral administration (63).

The present study showed that as regards the pre-operative Bisphosphonate of the studied sample shows that 19(95.0%) had Pre-operative Bisphosphonate. Lab investigation of the studied sample show that 12(60.0%) had low Ca Vit D and High ALK Phosph. Preoperative Medications of the studied sample show that all patients take calcium vit D. Lab investigation of the studied sample shows that 6 (30.0%) had 4 months postoperative, 3(15%) had 3 months postoperative and 10(50%) had 6 months postoperative.

Our results were supported by the study of Ruck et al.(36), as they reported that fifty-nine children (from 60) were receiving pamidronate treatment, a form of bisphosphonates, and started this treatment at a mean age of 1 year and 9 months, SD: 2 years and 1 month, with the youngest child starting pamidronate treatment at 8 days of age. The other child was using another type of bisphosphonate treatment, zoledronate, and started this treatment at 3 years and 7 months.

Similarly, Sterian et al.(87) demonstrated that prior to the surgical intervention, patients had a bisphosphonate treatment for 7 days.

Moreover, Langlais et al.,(102) revealed that all patients received intravenous bisphosphonates preoperatively.

A better quality of life including improved mobility and functional independence are the main goals of treatment for children with OI. These therapeutic plans should be based on a long-term multidisciplinary approach, which includes medical treatment with bisphosphonates, orthopedic treatment for fractures and deformity correction and rehabilitation (87).

The benefits of a telescoping intramedullary rod in fractures and deformity of long bones in children with OI are well known. The major and unsolved inconvenience of any telescopic system design is the lack of rotational stability. In children with OI, this problem can be associated with insufficient longitudinal bone stability (in the case of shortening of a segment at surgery or due to weakness of bone tissue) and diminished healing capacity. Furthermore, all telescoping systems are not implants for immediate weight-bearing. Only when radiological evidence of callus formation is present can active physiotherapy and weight-bearing with the aid of orthoses be started. In children with severe forms of OI, the long bones are narrow and often not suitable for telescoping rods. In such a situation, regular or elastic nailing achieves the required outcomes. (86).

The current study shows that functional score of the studied sample shows that the highest functional score frequency was 2 to 5 and 3 to 6 (15% and 15% respectively). Radiological scores show that the majority had a score of11 (95.0%).

Our results were supported by the study of Günay et al.,(103) as they reported that in all cases, it was observed that there was improvement in the deformities after the operation. The radiological and clinical union was achieved in all of the bones.

In the study of Popkov,,(104) radiographs demonstrated bone union in the femur 46 days after surgery. The fixator was removed under GA. Radiographic evaluations of angles at the right side demonstrated an mLDFA-93°; and mMPTA-87°. An orthotic was used after fixator removal and maintained for 3 weeks. At the follow-up visit 9 months after fixator removal, clinical alignment remained excellent without any recurrence of deformity. Bone remodeling with restitution of the medullary canal was noted on the radiographs. Radiographic evaluations of angles on the right side were: mLDFA-94°; mMPTA-92°; and mLDTA-84°. The values were close to the ones measured after fixator removal. Telescoping of the intramedullary nails indicated longitudinal growing of the femur. The patient was able to stand and work with an aide or walker and without pain. The range of motion in the hip and knee joints was not restricted. Bisphosphonate treatment had been resumed at that moment. At the follow-up visit 17 months after fixator removal, there was no decrease in functional abilities. At 1.5 years postoperatively, the FAQ ((Gillette Functional Assessment Questionnaire Ambulation Scale (FAQ)) score was 6.

Also, Sterian et al.,(87) reported that the first surgical procedure was made at the age of 4 years and 3 months when a Kirschner wire was used to stabilize the left femur after multiple corrective osteotomies and cast immobilization, procedure that had a poor outcome as the wire slipped after 3 weeks destabilizing the osteotomies and putting the soft tissue at risk. After this episode, a revision surgery was carried out to remove the wire and replace it with a Rush nail, which proved to have good results until the age of 5 when the distal end of the rod punctured the cortical bone of the femur and produced severe discomfort and eventually got replaced by a larger Rush nail.

Furthermore, Ruck et al.(36), indicated that most children obtained at least 90° AROM (Rehabilitation consisted of active range of motion) in the flexion of both hips and knees at 5 weeks post-initial FD (The Fassier-Duval) rodding of the femora. Twelve out of 40 had less than 90° of left knee flexion; seven out of 40 had a minimum of 80°. Ninety degrees of knee flexion is needed to climb and descend stairs alternately. Their findings indicate that, following the removal of the back slabs and 5 days of rehabilitation, a large majority of the children regained AROM ≥90° of the knees and hips. Their experience suggests that the absence of a knee arthrotomy in the FD rodding system favors this high degree of AROM 5 weeks after surgery.

In addition, Persiani et al.,(101) revealed that the osteosynthesis with the FD telescopic nail, performed with the minimally invasive surgical technique, has improved the management of deformities in OI.

The main advantage with the Fassier Duval system is that all the maneuvers for placing the components require no arthrotomy and no joint damage. This telescopic rod achieves this by allawing the operator to insert the components in the distal epiphysis under Rx control so that the growth plate takes minimal damage, and the joint surface is protected (36).

ELIGIBILITY:
Inclusion Criteria:

* Growing child (3-12 ys) Bony deformities with other symptoms and signs of OI

Exclusion Criteria:

* Old age (post Physeal closure). Other causes of bone deformities rather than OI

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Radiological score | During one year
  Bone union, callus formation, remodeling and fracture line

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided